CLINICAL TRIAL: NCT05986357
Title: The Relation Between Maternal Serum High Sensitivity C Reactive Protein and Total and Differential Leucocytic Count Levels in Healthy Pregnant Women With Threatened Abortion and the Outcome of Pregnancy
Brief Title: The Relation of High Sensitivity C Reactive Protein and Total Leucocytic Count Levels in Threatened Abortion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Other Study IDs: C reactive protein abortion
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Abortion Early
Keywords: C reactive protein; total and differential leucocytic count; abortion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: 120 healthy women presenting with threatened miscarriage.
  Interventions: Diagnostic Test: maternal serum C reactive protein; Diagnostic Test: total leucocytic count levels; Diagnostic Test: differential leucocytic count levels
- Control group: 120 healthy women with an uncomplicated single pregnancy.
  Interventions: Diagnostic Test: maternal serum C reactive protein; Diagnostic Test: total leucocytic count levels; Diagnostic Test: differential leucocytic count levels

INTERVENTIONS:
Diagnostic Test: maternal serum C reactive protein — maternal serum high sensitivity C reactive protein
Diagnostic Test: total leucocytic count levels — total leucocytic count levels
Diagnostic Test: differential leucocytic count levels — differential leucocytic count levels

SUMMARY:
to identify the relation between maternal serum high sensitivity C reactive protein and total and differential leucocytic count values in healthy pregnant women with threatened abortion and the outcome of pregnancy

DETAILED DESCRIPTION:
observational prospective cohort research will be pregnant women attending to obstetrics and gynecology department of University Hospital. After enrollment, participants will be divided into two groups:

* Study group: had 120 healthy women presenting with threatened miscarriage.
* Control group: had 120 healthy women with an uncomplicated single pregnancy. informed permission will be obtained. All cases subjected to the following: taking complete history, General examination, Special investigations including Obstetric ultrasonography for assessment of gestational age, and exclusion of congenital anomalies or multi-fetal gestation. Laboratory investigations including Estimation of the complete blood picture (CBC), Highly sensitive CRP (HS-CRP) single measurement, Women over 1st trimester abdominal ultrasonographic examination (6-13weeks) using Toshiba with transabdominal transducer probe frequency of 7 MHz to evaluate the following data: Measuring of the fetal crown-rump length (CRL) done to confirm the fetal gestational age and the viability of the fetus. Gestational age will be calculated from the beginning of the last regular menstrual cycle. Women who had hormone therapy or progesterone supplements, as well as pregnancies with a discrepancy between LMP and crown rump length of more than three days, were excluded from the research.

Pregnant women will be under close follow up every 2 weeks by: Obstetric U/S, Measure blood pressure and inform us if severe bleeding occurs.

ELIGIBILITY:
Inclusion Criteria:

* Single intrauterine pregnancy with vaginal hemorrhage and/or abdominal pain in the study group,
* an ultrasound showing an intrauterine gestational sac with a live fetus and a regular fetal heartbeat, with/without a sub-chorionic hematoma,
* healthy women who come for routine antenatal care with spontaneous pregnancy.

Exclusion Criteria:

* Age over 40
* smoking
* multiple pregnancies
* endocrinological diseases
* history of repeated spontaneous abortions.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Single intrauterine pregnancy with vaginal hemorrhage and/or abdominal pain in the study group, an ultrasound showing an intrauterine gestational sac with a live fetus and a regular fetal heartbeat, with/without a sub-chorionic hematoma, and healthy women who come for routine antenatal care with spontaneous pregnancy.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Highly sensitive CRP (HS-CRP) | 9 months
  A high level of hs-CRP, i.e., greater than 3 mg/L,
total leucocytic count | 9 months
  measures the number of white blood cells (WBCs) in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided